CLINICAL TRIAL: NCT04749186
Title: Achieving Lumbar Epidural Block Competency in Inexperienced Trainees After a Structured Teaching Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: European e-Learning School in Obstetric Anesthesia (Other)
Collaborators: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EESOA9
Record Dates: First submitted 2021-02-04; First posted 2021-02-11 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2021-04

CONDITIONS: Educational Problems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Structured Didactic Model Group (Active Comparator): A standardized video lessons (anatomy and technique), construction of a 3D epidural plastic module, practical training by using an epidural simulator with the CompuFlo Trainer instrument, and practical training with the eye-tracking assisted technique.
  Interventions: Device: Compuflo Epidural Training Instrument
- Standard Training Model (No Intervention): The standard local institutional teaching program

INTERVENTIONS:
Device: Compuflo Epidural Training Instrument — The intervention will consist of a Structured Didactic Model. It will include the following: two standardized video lessons (anatomy and technique), construction of a 3D epidural plastic module, practical training by using an epidural simulator with the CompuFlo Trainer instrument, and practical training with the eye-tracking assisted technique.
  Other Names: Eye tracking glasses; Standardized educational videorecordings; Epidural Simulator
  Arms: Structured Didactic Model Group

SUMMARY:
There is currently no universally accepted, comprehensive, or standard systematic way to teach the epidural block. Typical teaching of epidural catheter placement consists of a combination of didactic education and hands-on experience, where apprentice and master approached the task together in the clinical setting, with live patients as the learning model.

The learning curve is one of the most common tools to assess how the physician in training is progressing at a skill, and it is defined as a curve generated by plotting the success or failure against the number of attempts. More complex learning curves using an acceptable and unacceptable failure rate can be constructed. To perform these more complex learning curves a statistical tool such as the Cumulative Sum Technique (CUSUM) may be used.

The CompuFlo Epidural Trainer can differentiate tissue types by pressure signatures that are imperceptible to touch. This allows the trainee to accurately identify the needle location and discriminate between false and true loss of resistance. Having displayed, recorded and printed a graph illustrating the procedure, may also lead to a greater appreciation of the anatomy of the structures the needle must pass.

Eye-tracking is the process of measuring either the point of gaze or the motion of an eye relative to the head. This method has been successfully used for proficiency assessment.

The aim of this study will be to investigate whether the use of a Structured Didactic Model (SDM) including standardized video lessons, construction of a 3D epidural module, practical training by using an epidural simulator with CompuFlo Trainer instrument, eye tracking assisted technique, may affect the CUSUM learning curve for lumbar epidural block in novice, inexperienced trainees and their eye-tracking patterns.

DETAILED DESCRIPTION:
Researchers will enroll 15 PGY3 trainees who have never performed an epidural block and are about to begin their obstetrics rotation. After having had the usual standard front-lecture on anatomy and technique, they will be randomized into two groups to receive (study group) or to not receive (control group) the additional SDM (Structured Didactic Model). The additional SDM will consist in two standardized video lessons (anatomy and technique), construction of a 3D epidural plastic module, practical training by using an epidural simulator with the CompuFlo Trainer instrument, and practical training with the eye-tracking assisted technique.

After the randomization and before their practice on the patients, all the trainees will undergo eye-tracking measurement of their visual patterns while performing the epidural block on an epidural simulator.

All trainees will perform lumbar epidural anesthesia under the supervision of their instructors in accordance with local Institutional policy and practice, with the standard routine equipment and monitoring. Every time the trainee will perform an epidural technique, the number of attempts, needle redirections, and effectiveness of the epidural block will be noted and used to construct the corresponding CUSUM curve.

When enough epidurals will be performed by each trainee to reach competence according to the CUSUM curve, a post hoc Power Analysis will be carried out to verify the 95% significance level and the 80 % test power. To study and compare the evolution of the success rate in each group a linear regression model will be applied.

ELIGIBILITY:
Inclusion Criteria:

* PGY3 trainees who have never performed an epidural block

Exclusion Criteria:

* PGY3 trainees who have already performed an epidural block

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
number of attempts | immediately after the procedure
  Every time the trainee will perform an epidural technique, a number of attempts will be noted and used to construct the corresponding CUSUM learning curve.
number of needle redirections | immediately after the procedure
  Every time the trainee will perform an epidural technique, a number of needle redirections will be noted and used to construct the corresponding CUSUM learning curve.
efficacy of epidural block | 20 minutes after the epidural procedure
  The efficacy of the epidural block will be evaluated by using a visual analogue pain scale where 0=no pain-100=worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Capogna, MD, Study Director — European e-Learning School in Obstetric Anesthesia
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No